CLINICAL TRIAL: NCT04753697
Title: A Phase 3, Multicenter, Multinational, Randomized, Double-Blind, Placebo-Controlled Induction and Maintenance Study to Evaluate the Efficacy and Safety of CC-93538 in Adult and Adolescent Subjects With Eosinophilic Esophagitis
Brief Title: A Study to Evaluate the Efficacy and Safety of CC-93538 in Adult and Adolescent Participants With Eosinophilic Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-93538-EE-001; U1111-1263-4351 (Registry Identifier: WHO); 2020-004336-16 (EudraCT Number)
Record Dates: First submitted 2021-02-05; First posted 2021-02-15 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; CC-93538; RPC4046; Adult; Adolescent; Gastrointestinal Diseases; Esophagitis; Gastroenteritis; Eosinophils; Eosinophilia; Esophageal Diseases; Allergic Diseases; Antibody, Monoclonal; Hypersensitivity; Immunologic factors; Physiological Effects of Drugs; cendakimab
MeSH Terms: conditions — Eosinophilic Esophagitis; Gastrointestinal Diseases; Esophagitis; Gastroenteritis; Eosinophilia; Esophageal Diseases; Hypersensitivity | interventions — cendakimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Administration of CC-93538 (Experimental): CC-93538 360 mg Subcutaneously (SC) once weekly for 24 weeks followed by CC-93538 360 mg SC once weekly for 24 weeks
  Interventions: Drug: CC-93538
- Administration of CC-93538 and Placebo (Experimental): CC-93538 360 mg SC once weekly for 24 weeks followed by CC-93538 360 mg SC once every other week for 24 weeks.
  During the Maintenance Phase, matching placebo will be administered once every other week on alternate weeks to maintain the blind.
  Interventions: Drug: CC-93538; Other: Placebo
- Administration of Placebo (Placebo Comparator): Matching placebo SC once weekly for 24 weeks followed by matching placebo SC once weekly for 24 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CC-93538 — Subcutaneous
  Other Names: RPC4046
  Arms: Administration of CC-93538; Administration of CC-93538 and Placebo
Other: Placebo — Subcutaneous
  Arms: Administration of CC-93538 and Placebo; Administration of Placebo

SUMMARY:
Study CC-93538-EE-001 is a Phase 3, multicenter, multinational, randomized, double-blind, placebo-controlled induction and maintenance study to evaluate the efficacy and safety of CC- 93538 in adult and adolescent participants with eosinophilic esophagitis (EoE). The study will incorporate a 24-week Induction Phase followed by a 24-week Maintenance Phase.

Participants will be randomized at the beginning of the study into 3 treatment arms:

* Placebo for Induction and Maintenance
* CC-93538 360 mg Subcutaneous (SC) once weekly for Induction followed by 360 mg SC once every other week for Maintenance
* CC-93538 360 mg SC once weekly for Induction and Maintenance

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy the following criteria to be enrolled in the study:

1. Male or female patients aged ≥ 12 and ≤ 75 years, with a body weight of > 40 kg.
2. Histologic evidence of eosinophilic esophagitis, defined as a peak count of ≥ 15 eosinophils/high-power field at 2 levels of the esophagus.

3 Participant-reported history of 4 or more Dysphagia Days within 2 consecutive weeks prior to end of screening.

4. Lack of complete response to an adequate trial of proton pump inhibitor (8 weeks). Participants on a proton pump inhibitor must have been on a stable dose for at least 4 weeks prior to first Screening Visit and agree to continue the same dose throughout the study.

5. Participants currently receiving inhaled corticosteroids, leukotriene receptor antagonists, or mast cell stabilizers for indications other than EoE, or medium potency topical corticosteroids for dermatologic conditions, must maintain stable doses for at least 4 weeks prior to the first Screening Visit and throughout the duration of the study.

6. Participants must agree to maintain a stable diet (including any food elimination diet for the treatment of food allergy or eosinophilic esophagitis) and not introduce any changes in their diet from the first Screening Visit to the end of the study.

7. Females of childbearing potential must have 2 negative pregnancy tests as verified by the Investigator prior to starting study therapy and agree to practice a highly effective method of contraception until 5 months after the last dose.

Exclusion Criteria:

The presence of any of the following will exclude a participant from enrollment:

1. Clinical or endoscopic evidence of other diseases that may affect the histologic, endoscopic, and clinical symptom evaluation for this study.
2. Other gastrointestinal disorders such as active Helicobacter pylori infection, esophageal varices, gastritis, colitis, celiac disease, Mendelian disorder associated with eosinophilic esophagitis, liver function impairment, or a known hereditary fructose intolerance.
3. Evidence of a severe endoscopic structural abnormality in the esophagus.
4. Esophageal dilation for symptom relief within 8 weeks prior to first Screening Visit or during the Screening Period, or if esophageal dilation is anticipated within 48 weeks of dosing during the study.
5. Evidence of immunosuppression, or of having received systemic immunosuppressive or immunomodulating drugs within 5 drug half-lives prior to the first Screening Visit.
6. Treatment with a high potency topical corticosteroid for dermatologic use, or a systemic corticosteroid within 8 weeks of the first Screening Visit.
7. Treatment with a swallowed topical corticosteroid, leukotriene receptor antagonist, or mast cell stabilizer for EoE, within 4 weeks of the first Screening Visit.
8. Treatment with oral or sublingual immunotherapy within 6 months of the first Screening Visit (any use will be prohibited during the study). Subcutaneous immunotherapy may be allowed if on stable doses for at least 3 months prior to the first Screening Visit and during the study.
9. Actively successful dietary modification adherence (e.g. food elimination diet), resulting in a complete response to EoE.
10. Prior treatment with CC-93538 during a Phase 1 or 2 clinical study.
11. Receipt of a live attenuated vaccine within 4 weeks of the first Screening Visit.
12. Any disease that would affect the conduct of the protocol or interpretation of the study results, or would put a patient at risk by participating in the study (e.g. severe uncontrolled asthma, infection causing eosinophilia, hypereosinophilic syndrome, or cardiovascular condition, or neurologic disorder or psychiatric illness that compromises the Participant's ability to accurately document symptoms of eosinophilic esophagitis).
13. Active or ongoing infections including parasitic/helminthic, hepatitis, tuberculosis, or human immunodeficiency virus.
14. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 4 weeks of the first Screening Visit.
15. Females who are pregnant or lactating.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (212):
- United States (115):
  - Local Institution - 144, Birmingham, Alabama
  - Local Institution - 158, Tuscaloosa, Alabama
  - Local Institution - 082, Phoenix, Arizona
  - Local Institution - 147, Phoenix, Arizona
  - Local Institution - 041, Scottsdale, Arizona
  - Local Institution - 029, Tucson, Arizona
  - Local Institution - 165, North Little Rock, Arkansas
  - Local Institution - 075, Lancaster, California
  - Local Institution - 047, Los Angeles, California
  - Local Institution - 084, Oakland, California
  - Local Institution - 160, San Diego, California
  - Local Institution - 068, Aurora, Colorado
  - Local Institution - 067, Colorado Springs, Colorado
  - Local Institution - 092, Denver, Colorado
  - Local Institution - 170, Littleton, Colorado
  - Local Institution - 128, Wheat Ridge, Colorado
  - Local Institution - 101, Bristol, Connecticut
  - Local Institution - 076, Farmington, Connecticut
  - Local Institution - 156, Hamden, Connecticut
  - Local Institution - 099, Clearwater, Florida
  - Local Institution - 036, Inverness, Florida
  - Local Institution - 042, Jacksonville, Florida
  - Local Institution - 161, Miami, Florida
  - Local Institution - 138, Miami, Florida
  - Local Institution - 110, North Miami Beach, Florida
  - Local Institution - 146, Orlando, Florida
  - Local Institution - 088, Orlando, Florida
  - Local Institution - 133, Orlando, Florida
  - Local Institution - 169, Pinellas Park, Florida
  - Local Institution - 168, Plantation, Florida
  - Local Institution - 037, Port Orange, Florida
  - Local Institution - 140, Sweetwater, Florida
  - Local Institution - 043, Atlanta, Georgia
  - Local Institution - 171, Atlanta, Georgia
  - Local Institution - 054, Atlanta, Georgia
  - Local Institution - 117, Macon, Georgia
  - Local Institution - 024, Idaho Falls, Idaho
  - Local Institution - 039, Chicago, Illinois
  - Local Institution - 167, Gurnee, Illinois
  - Local Institution - 118, Indianapolis, Indiana
  - Local Institution - 127, Clive, Iowa
  - Local Institution - 094, Iowa City, Iowa
  - Local Institution - 035, Kansas City, Kansas
  - Local Institution - 046, Florence, Kentucky
  - Local Institution - 019, Louisville, Kentucky
  - Local Institution - 003, Baton Rouge, Louisiana
  - Local Institution - 020, Metairie, Louisiana
  - Local Institution - 044, Metairie, Louisiana
  - Local Institution - 109, Baltimore, Maryland
  - Local Institution - 065, Catonsville, Maryland
  - Local Institution - 164, Columbia, Maryland
  - Local Institution - 070, Glen Burnie, Maryland
  - Local Institution - 012, Hagerstown, Maryland
  - Local Institution - 053, Boston, Massachusetts
  - Local Institution - 097, Boston, Massachusetts
  - Local Institution - 017, Framingham, Massachusetts
  - Local Institution - 083, South Dartmouth, Massachusetts
  - Local Institution - 081, Springfield, Massachusetts
  - Local Institution - 009, Worcester, Massachusetts
  - Local Institution - 098, Troy, Michigan
  - Local Institution - 014, Wyoming, Michigan
  - Local Institution - 115, Plymouth, Minnesota
  - Local Institution - 049, Rochester, Minnesota
  - Local Institution - 034, Flowood, Mississippi
  - Local Institution - 007, Kansas City, Missouri
  - Local Institution - 032, St Louis, Missouri
  - Local Institution - 038, Omaha, Nebraska
  - Local Institution - 015, Lebanon, New Hampshire
  - Local Institution - 139, Albuquerque, New Mexico
  - Local Institution - 028, Great Neck, New York
  - Local Institution - 051, New York, New York
  - Local Institution - 154, New York, New York
  - Local Institution - 011, New York, New York
  - Local Institution - 116, Syracuse, New York
  - Local Institution - 142, Syracuse, New York
  - Local Institution - 016, Chapel Hill, North Carolina
  - Local Institution - 045, Charlotte, North Carolina
  - Local Institution - 106, Durham, North Carolina
  - Local Institution - 131, Greensboro, North Carolina
  - Local Institution - 126, Kinston, North Carolina
  - Local Institution - 130, Beavercreek, Ohio
  - Local Institution - 006, Cincinnati, Ohio
  - Local Institution - 001, Cincinnati, Ohio
  - Local Institution - 052, Cincinnati, Ohio
  - Local Institution - 072, Cleveland, Ohio
  - Local Institution - 145, Columbus, Ohio
  - Local Institution - 059, Columbus, Ohio
  - Local Institution - 166, Oklahoma City, Oklahoma
  - Local Institution - 120, Hershey, Pennsylvania
  - Local Institution - 025, Philadelphia, Pennsylvania
  - Local Institution - 155, Pottsville, Pennsylvania
  - Local Institution - 066, Providence, Rhode Island
  - Local Institution - 143, Anderson, South Carolina
  - Local Institution - 057, Greenville, South Carolina
  - Local Institution - 114, Chattanooga, Tennessee
  - Local Institution - 095, Nashville, Tennessee
  - Local Institution - 105, Cedar Park, Texas
  - Local Institution - 148, Dallas, Texas
  - Local Institution - 112, Houston, Texas
  - Local Institution - 079, Rockwell, Texas
  - Local Institution - 008, San Antonio, Texas
  - Local Institution - 077, Southlake, Texas
  - Local Institution - 104, Tyler, Texas
  - Local Institution - 157, Draper, Utah
  - Local Institution - 125, Ogden, Utah
  - Local Institution - 074, Salt Lake City, Utah
  - Local Institution - 027, Leesburg, Virginia
  - Local Institution - 013, Lynchburg, Virginia
  - Local Institution - 064, Richmond, Virginia
  - Local Institution - 134, Roanoke, Virginia
  - Local Institution - 137, Spokane, Washington
  - Local Institution - 023, Vancouver, Washington
  - Local Institution - 085, Milwaukee, Wisconsin
  - Local Institution - 060, Milwaukee, Wisconsin
  - Local Institution - 121, Casper, Wyoming
- Argentina (3):
  - Local Institution - 697, Buenos Aires
  - Local Institution - 695, Mar del Plata
  - Local Institution - 696, Quilmes
- Australia (14):
  - Local Institution - 548, Concord, New South Wales
  - Local Institution - 554, Liverpool, New South Wales
  - Local Institution - 540, Westmead, New South Wales
  - Local Institution - 546, Maroorchydore, Queensland
  - Local Institution - 550, South Brisbane, Queensland
  - Local Institution - 542, Woolloongabba, Queensland
  - Local Institution - 552, Adelaide, South Australia
  - Local Institution - 545, Elizabeth Vale, South Australia
  - Local Institution - 553, Clayton, Victoria
  - Local Institution - 543, Footscray, Victoria
  - Local Institution - 539, Melbourne, Victoria
  - Local Institution - 549, Murdoch, Western Australia
  - Local Institution - 538, Fitzroy
  - Local Institution - 547, Western Australia
- Austria (3):
  - Local Institution - 437, Burgenland
  - Local Institution - 434, Graz
  - Local Institution - 436, Linz
- Belgium (4):
  - Local Institution - 515, Brussels
  - Local Institution - 516, Kortrijk
  - Local Institution - 514, Leuven
  - Local Institution - 512, West-Vlaanderen
- Canada (7):
  - Local Institution - 201, Calgary, Alberta
  - Local Institution - 208, Edmonton, Alberta
  - Local Institution - 205, Edmonton, Alberta
  - Local Institution - 203, Vancouver, British Columbia
  - Local Institution - 206, Victoria, British Columbia
  - Local Institution - 207, Ottawa, Ontario
  - Local Institution - 200, Vaughan, Ontario
- Germany (8):
  - Local Institution - 330, Bayern
  - Local Institution - 332, Brandenburg
  - Local Institution - 339, Frankfurt am Main
  - Local Institution - 336, Hamburg
  - Local Institution - 333, Leipzig
  - Local Institution - 338, Leipzig
  - Local Institution - 340, München
  - Local Institution - 337, München
- Israel (6):
  - Local Institution - 281, Haifa
  - Local Institution - 283, Holon
  - Local Institution - 280, Jerusalem
  - Local Institution - 282, Jerusalem
  - Local Institution - 278, Tel Aviv
  - Local Institution - 279, Ẕerifin
- Italy (5):
  - Local Institution - 257, Genova
  - Local Institution - 254, Milan
  - Local Institution - 255, Padua
  - Local Institution - 252, Pisa
  - Local Institution - 253, Rome
- Japan (17):
  - Local Institution - 600, Nishinomiya, Hyōgo
  - Local Institution - 595, Bunkyo-ku, Tokyo
  - Local Institution - 599, Setagaya-ku, Tokyo
  - Local Institution - 593, Akita
  - Local Institution - 606, Isehara City, Kanagawa
  - Local Institution - 597, Kobe
  - Local Institution - 598, Maebashi
  - Local Institution - 604, Nagoya
  - Local Institution - 607, Nagoya
  - Local Institution - 592, Niigata
  - Local Institution - 603, Okayama
  - Local Institution - 591, Osaka
  - Local Institution - 601, Shibukawa
  - Local Institution - 602, Shinjuku-Ku
  - Local Institution - 605, Tokyo
  - Local Institution - 596, Toyoake
  - Local Institution - 590, Yamagata
- Poland (11):
  - Local Institution - 385, Bydgoszcz
  - Local Institution - 389, Częstochowa
  - Local Institution - 390, Gdansk
  - Local Institution - 388, Katowice
  - Local Institution - 392, Lódz
  - Local Institution - 387, Warsaw
  - Local Institution - 393, Warsaw
  - Local Institution - 383, Warsaw
  - Local Institution - 391, Wroclaw
  - Local Institution - 386, Wroclaw
  - Local Institution - 384, Wroclaw
- Portugal (4):
  - Local Institution - 307, Lisbon
  - Local Institution - 305, Lisbon
  - Local Institution - 306, Porto
  - Local Institution - 308, Porto
- Spain (6):
  - Local Institution - 408, Barcelona
  - Local Institution - 410, Córdoba
  - Local Institution - 409, Madrid
  - Local Institution - 413, Madrid
  - Local Institution - 411, Marbella
  - Local Institution - 412, Seville
- Local Institution - 357, Lausanne, Switzerland
- United Kingdom (8):
  - Local Institution - 228, Belfast Northern Ireland
  - Local Institution - 231, Birmingham
  - Local Institution - 234, Cardiff
  - Local Institution - 235, Chorley
  - Local Institution - 233, Hexam
  - Local Institution - 236, Liverpool
  - Local Institution - 237, Manchester
  - Local Institution - 226, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- [Derived] Dellon ES, Charriez CM, Zhang S, Falk GW, Oliva S, Ma C, Siffledeen J, Schroeder S, Philpott H, Vanuytsel T, Abe Y, Li K, Zema CL, Venkatasamy A, Yeshokumar AK, Oh YS, Schoepfer A. Cendakimab in Adults and Adolescents with Eosinophilic Esophagitis. NEJM Evid. 2025 Oct;4(10):EVIDoa2500095. doi: 10.1056/EVIDoa2500095. Epub 2025 Sep 23. PMID 40985784
- [Derived] Charriez CM, Zhang S, de Oliveira CHMC, Patel V, Oh YS, Hirano I, Schoepfer A, Dellon ES. Design of a phase 3, randomized, double-blind, placebo-controlled, 48-week study to evaluate the efficacy and safety of cendakimab in adult and adolescent patients with eosinophilic esophagitis. Contemp Clin Trials. 2024 Dec;147:107708. doi: 10.1016/j.cct.2024.107708. Epub 2024 Oct 9. PMID 39384067
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/home

RESULTS

PARTICIPANT FLOW:
Groups:
- CC-93538 360 mg QW: Participants with Eosinophilic Esophagitis received 360 mg CC-93538 SC once every week in the 24-week induction phase followed by 24-week maintenance phase.
- CC-93538 360 mg QW/Q2W: Participants with Eosinophilic Esophagitis received 360 mg CC-93538 SC once in a week (QW) in the 24-week induction phase and once every other week in 24-week maintenance phase.
- Placebo: Participants with active eosinophilic esophagitis received CC-93538 matching placebo during 24-week induction phase followed by 24-week maintenance phase.
Period: Pre-Treatment Period
Arm/Group | CC-93538 360 mg QW | CC-93538 360 mg QW/Q2W | Placebo
Started (The Intent-to-Treat (ITT)population consist of all randomized participants and analyzed according to their randomized treatment group regardless of whether or not the participants received CC-93538 or placebo.) | 143 | 143 | 144
Completed | 143 | 141 | 143
Not Completed | 0 | 2 | 1
Period: Induction Phase
Arm/Group | CC-93538 360 mg QW | CC-93538 360 mg QW/Q2W | Placebo
Started | 143 | 141 | 143
Completed | 127 | 134 | 136
Not Completed | 16 | 7 | 7
Not completed — Withdrawal by Subject | 12 | 5 | 6
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0
Period: Maintenance Phase
Arm/Group | CC-93538 360 mg QW | CC-93538 360 mg QW/Q2W | Placebo
Started | 114 (13 participants who completed induction phase did not enter maintenance phase) | 117 (17 participants who completed induction phase did not enter maintenance phase) | 90 (46 participants who completed induction phase did not enter maintenance phase)
Completed | 107 | 110 | 82
Not Completed | 7 | 7 | 8
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 4 | 6
Not completed — Lost to Follow-up | 2 | 2 | 0
Not completed — NON-COMPLIANCE WITH STUDY DRUG | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1
Not completed — WITHDRAWAL BY PARENT/GUARDIAN | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CC-93538 360 mg QW | CC-93538 360 mg QW/Q2W | Placebo | Total
Number analyzed (Participants) | 143 | 143 | 144 | 430
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (11.79) | 34.8 (12.24) | 36.2 (12.16) | 35.6 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 33 | 45 | 131
  Male | 90 | 110 | 99 | 299
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 6 | 17
  Not Hispanic or Latino | 135 | 138 | 137 | 410
  Unknown or Not Reported | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 5 | 10 | 11 | 26
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 2 | 3 | 0 | 5
  White | 134 | 128 | 130 | 392
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Dysphagia Days (DD) at Week 24
Description: Dysphagia Days (DD) was assessed using a modified daily symptom diary (mDSD). The DD was evaluated over the prior 14-day period using the mDSD, which includes 6 primary questions. These questions assess solid food consumption that day (Q1), experience with trouble swallowing (Q2), food going down slowly (Q3), food getting stuck in the throat or chest (Q4), actions taken by participants to obtain relief (Q5), and any pain associated with swallowing (Q6). The number of DD was normalized by calculating the number of diary days with a "yes" to any or all of Q2, Q3, and Q4 in the 14-day period prior to a visit, dividing by the number of measurable diary days in the 14-day period, and then multiplying by the length of the period (14). A measurable diary day for DD is defined as a diary day for which Questions 2 to 4 are answered. Mean DD ranges from 0 to 14 for the 14-day period.
Time Frame: Baseline (Day 1) and Week 24
Population: The Intent-to-Treat (ITT) population consist of all randomized participants and analyzed according to their randomized treatment group regardless of whether or not the participant received IP CC-93538 or placebo. Number of participants with observed values at the specified timepoint are included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Induction Phase - CC-93538 360 mg QW: Participants with Eosinophilic Esophagitis received 360 mg CC-93538 SC once every week in the 24-week induction phase.
- Induction Phase - Placebo: Participants with Eosinophilic Esophagitis received 360 mg CC-93538 matching placebo SC once every week in the 24-week induction phase.
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo
Number analyzed (Participants) | 236 | 124
days | -6.85 (5.259) | -4.98 (5.075)
Statistical Analysis 1: Comparison: Induction Phase - CC-93538 360 mg QW vs Induction Phase - Placebo; Test type: Superiority; p = 0.0005, ANCOVA; Difference in Least Square Mean = -1.91, 95% CI 2-sided [-2.97 to -0.84], Standard Error of Mean 0.544

2. Primary Outcome: Percentage of Participants With Peak Esophageal Eosinophil Count <= 6/High-power Field (Hpf) at Week 24
Description: Blood samples were collected to assess esophageal eosinophil count.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Induction Phase - CC-93538 360 mg QW: Participants with Eosinophilic Esophagitis received 360 mg CC-93538 SC once every week in the 24 week induction phase.
- Induction Phase - Placebo: Participants with Eosinophilic Esophagitis received 360 mg CC-93538 matching placebo SC once every week in the 24 week induction phase.
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo
Number analyzed (Participants) | 249 | 129
percentage of participants | 34.1 | 3.1
Statistical Analysis 1: Comparison: Induction Phase - CC-93538 360 mg QW vs Induction Phase - Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Imputed data is used in CMH test, which is stratified by Steroid Inadequate Responder/Intolerant status; Difference in percentage = 26.4, 95% CI 2-sided [20.6 to 32.2]

3. Secondary Outcome: Percentage of Participants With Peak Esophageal Eosinophil Count <= 6/High-power Field (Hpf) at Week 48
Description: Blood samples were collected to assess esophageal eosinophil count.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Maintenance Phase - CC-93538 360 mg QW: Participants with Eosinophilic Esophagitis received 360 mg CC-93538 SC once every week in the 24 week maintenance phase.
- Maintenance Phase - CC-93538 360 mg Q2W: Participants with Eosinophilic Esophagitis received 360 mg CC-93538 SC once every other week in the 24 week maintenance phase.
- Maintenance Phase - Placebo: Participants with Eosinophilic Esophagitis received 360 mg CC-93538 matching placebo SC once every week in the 24 week maintenance phase.
Arm/Group | Maintenance Phase - CC-93538 360 mg QW | Maintenance Phase - CC-93538 360 mg Q2W | Maintenance Phase - Placebo
Number analyzed (Participants) | 104 | 108 | 82
percentage of participants | 37.5 | 34.3 | 4.9
Statistical Analysis 1: Comparison: Maintenance Phase - CC-93538 360 mg QW vs Maintenance Phase - Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Imputed data is used in CMH test, which is stratified by Steroid Inadequate Responder/Intolerant status; DIFFERENCE IN RESPONSE RATE AFTER MI(%) = 18.4, 95% CI 2-sided [11.3 to 25.5]
Statistical Analysis 2: Comparison: Maintenance Phase - CC-93538 360 mg Q2W vs Maintenance Phase - Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Imputed data is used in CMH test, which is stratified by Steroid Inadequate Responder/Intolerant status; DIFFERENCE IN RESPONSE RATE AFTER MI(%) = 17.0, 95% CI 2-sided [10.1 to 24.0]

4. Secondary Outcome: Percentage of Participants With Peak Esophageal Eosinophil Count < 15/High-power Field (Hpf) at Week 24
Description: Blood samples were collected to assess esophageal eosinophil count.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo
Number analyzed (Participants) | 249 | 129
percentage of participants | 53.0 | 4.7
Statistical Analysis 1: Comparison: Induction Phase - CC-93538 360 mg QW vs Induction Phase - Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Imputed data is used in CMH test, which is stratified by Steroid Inadequate Responder/Intolerant status; DIFFERENCE IN RESPONSE RATE AFTER MI (%) = 40.0, 95% CI 2-sided [33.3 to 46.7]

5. Secondary Outcome: Percentage of Participants With Peak Esophageal Eosinophil Count < 15/High-power Field (Hpf) at Week 48
Description: Blood samples were collected to assess esophageal eosinophil count.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance Phase - CC-93538 360 mg QW | Maintenance Phase - CC-93538 360 mg Q2W | Maintenance Phase - Placebo
Number analyzed (Participants) | 104 | 108 | 82
percentage of participants | 50.0 | 50.0 | 8.5
Statistical Analysis 1: Comparison: Maintenance Phase - CC-93538 360 mg QW vs Maintenance Phase - Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Imputed data is used for all in CMH test, which is stratified by Steroid Inadequate Responder/Intolerant status; DIFFERENCE IN RESPONSE RATE AFTER MI (%) = 25.7, 95% CI 2-sided [17.8 to 33.6]
Statistical Analysis 2: Comparison: Maintenance Phase - CC-93538 360 mg QW vs Maintenance Phase - Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Imputed data is used for all in CMH test, which is stratified by Steroid Inadequate Responder/Intolerant status; DIFFERENCE IN RESPONSE RATE AFTER MI (%) = 27.7, 95% CI 2-sided [19.7 to 35.7]

6. Secondary Outcome: Change From Baseline in Mean Dysphagia Days (DD) at Week 48
Description: as for outcome 1
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Maintenance Phase - CC-93538 360 mg QW | Maintenance Phase - CC-93538 360 mg Q2W | Maintenance Phase - Placebo
Number analyzed (Participants) | 100 | 101 | 75
days | -7.71 (5.401) | -8.07 (5.292) | -6.20 (5.118)
Statistical Analysis 1: Comparison: Maintenance Phase - CC-93538 360 mg QW vs Maintenance Phase - Placebo; Test type: Superiority; p = 0.0006, ANCOVA; DIFFERENCE IN LSM = -2.26, 95% CI 2-sided [-3.55 to -0.98], Standard Error of Mean 0.655
Statistical Analysis 2: Comparison: Maintenance Phase - CC-93538 360 mg QW vs Maintenance Phase - Placebo; Test type: Superiority; p = 0.0002, ANCOVA; DIFFERENCE IN LSM = -2.49, 95% CI [-3.78 to -1.20], Standard Error of Mean 0.657

7. Secondary Outcome: Change From Baseline in Eosinophilic Esophagitis (EoE) Endoscopic Reference Score (EREFS) at Week 24
Description: The EREFS, measures features of EoE including esophageal edema, fixed rings, exudates, furrows, and strictures. The instrument grades edema as none (0) or present (1) or severe; furrows as absent (0), present (1); rings as none (0), mild (1), moderate (2) and severe (3); exudates as none (0), mild (1) or severe (2); and strictures as absent (0) or present (1). Two sub-component scores will be calculated by adding up the grade from respective features across the 3 esophagus levels (proximal, mid, and distal). Inflammation composite score (ranging 0 to 12) includes edema, furrows and exudates while remodeling composite score (0 to 12) consist of stricture and fixed rings. The EREFS total score is the sum of the inflammation and remodeling composite scores. The EREFS total score ranges from 0 to 24. High score signifies severe condition.
Time Frame: Baseline (Day 1) , Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo
Number analyzed (Participants) | 249 | 128
score on a scale | -6.0 (4.54) | -1.5 (4.26)
Statistical Analysis 1: Comparison: Induction Phase - CC-93538 360 mg QW vs Induction Phase - Placebo; Test type: Superiority; p < 0.0001, ANCOVA; DIFFERENCE IN LSM = -4.0, 95% CI 2-sided [-4.8 to -3.2], Standard Error of Mean 0.42

8. Secondary Outcome: Change From Baseline in Eosinophilic Esophagitis (EoE) Endoscopic Reference Score (EREFS) at Week 48
Description: as for outcome 7
Time Frame: Baseline (Day 1) , Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Maintenance Phase - CC-93538 360 mg QW | Maintenance Phase - CC-93538 360 mg Q2W | Maintenance Phase - Placebo
Number analyzed (Participants) | 103 | 105 | 79
score on a scale | -6.6 (4.24) | -6.5 (4.57) | -3.2 (4.15)
Statistical Analysis 1: Comparison: Maintenance Phase - CC-93538 360 mg QW vs Maintenance Phase - Placebo; Test type: Superiority; p < 0.0001, ANCOVA; DIFFERENCE IN LSM = -3.5, 95% CI 2-sided [-4.5 to -2.4], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: Maintenance Phase - CC-93538 360 mg QW vs Maintenance Phase - Placebo; Test type: Superiority; p < 0.0001, ANCOVA; DIFFERENCE IN LSM = -3.1, 95% CI 2-sided [-4.1 to -2.1], Standard Error of Mean 0.51

9. Secondary Outcome: Change From Baseline in Mean Adjusted Eosinophilic Esophagitis Histology Scoring System (EoEHSS) Grade Score at Week 24
Description: EoEHSS evaluates the grade (severity) of multiple pathologic features in esophageal biopsies. It has 8 features eosinophil inflammation, basal zone hyperplasia, eosinophil abscess, eosinophil surface layering, dilated intercellular spaces, surface epithelial alteration, dyskeratotic epithelial cells, and lamina propria fibrosis. In 3 separate esophagus levels (proximal, mid, and distal), each feature is scored independently for grade using a 4-point Likert scale (0 [absent] to 3 [severe]). The mean adjusted grade score is calculated by averaging the adjusted scores for the 3 levels (proximal, mid, and distal). The mean adjusted scores range from 0 to 100. High score signifies severe condition.
Time Frame: Baseline (Day 1), Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo
Number analyzed (Participants) | 249 | 129
Score on a scale | -30.20 (15.811) | -6.47 (15.755)
Statistical Analysis 1: Comparison: Induction Phase - CC-93538 360 mg QW vs Induction Phase - Placebo; Test type: Superiority; p < 0.0001, ANCOVA; DIFFERENCE IN LSM = -22.51, 95% CI 2-sided [-25.50 to -19.51], Standard Error of Mean 1.528

10. Secondary Outcome: Change From Baseline in Mean Adjusted Eosinophilic Esophagitis Histology Scoring System (EoEHSS) Grade Score at Week 48
Description: as for outcome 9
Time Frame: Baseline (Day 1) , Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Maintenance Phase - CC-93538 360 mg QW | Maintenance Phase - CC-93538 360 mg Q2W | Maintenance Phase - Placebo
Number analyzed (Participants) | 104 | 108 | 82
score on a scale | -30.35 (17.146) | -30.96 (15.864) | -6.17 (16.579)
Statistical Analysis 1: Comparison: Maintenance Phase - CC-93538 360 mg QW vs Maintenance Phase - Placebo; Test type: Superiority; p < 0.0001, ANCOVA; DIFFERENCE IN LSM = -18.13, 95% CI 2-sided [-21.85 to -14.40], Standard Error of Mean 1.900
Statistical Analysis 2: Comparison: Maintenance Phase - CC-93538 360 mg Q2W vs Maintenance Phase - Placebo; Test type: Superiority; p < 0.0001, ANCOVA; DIFFERENCE IN LSM = -19.22, 95% CI 2-sided [-22.90 to -15.53], Standard Error of Mean 1.880

11. Secondary Outcome: Change From Baseline in Mean Adjusted Eosinophilic Esophagitis Histology Scoring System (EoEHSS) Stage Score at Week 24
Description: EoEHSS evaluates the stage (extent) of multiple pathologic features in esophageal biopsies. It has 8 features eosinophil inflammation (determined by peak EoS count(PEC)) and presence of basal zone hyperplasia, eosinophil abscess, eosinophil surface layering, dilated intercellular spaces, surface epithelial alteration, dyskeratotic epithelial cells, and lamina propria fibrosis in epithelium . In 3 separate esophagus levels (proximal, mid, and distal), each feature is scored independently for stage using a 4-point Likert scale (0 [absent], 1[PEC ≥15/hpf in <33% of hpfs or (any grade >0) <33% of epithelium for other features], 2 [PEC ≥15/hpf in 33-66% of hpfs or (any grade >0) in 33-66% of epithelium to 3 [PEC ≥15/hpf in >66% of hpfs or (any grade >0) in > 66% of epithelium]). The mean adjusted stage score is calculated by averaging the adjusted scores for the 3 levels (proximal, mid, and distal). The mean adjusted scores range from 0 to 100. High score signifies severe condition.
Time Frame: Baseline (Day 1), Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo
Number analyzed (Participants) | 249 | 129
Score on a scale | -36.71 (19.370) | -9.90 (17.583)
Statistical Analysis 1: Comparison: Induction Phase - CC-93538 360 mg QW vs Induction Phase - Placebo; Test type: Superiority; p < 0.0001, ANCOVA; DIFFERENCE IN LSM = -25.40, 95% CI 2-sided [-28.92 to -21.89], Standard Error of Mean 1.793

12. Secondary Outcome: Change From Baseline in Mean Adjusted Eosinophilic Esophagitis Histology Scoring System (EoEHSS) Stage Score at Week 48
Description: as for outcome 11
Time Frame: Baseline (Day 1) , Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Maintenance Phase - CC-93538 360 mg QW | Maintenance Phase - CC-93538 360 mg Q2W | Maintenance Phase - Placebo
Number analyzed (Participants) | 104 | 108 | 82
score on a scale | -36.30 (20.904) | -37.36 (19.290) | -8.38 (19.935)
Statistical Analysis 1: Comparison: Maintenance Phase - CC-93538 360 mg QW vs Maintenance Phase - Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; DIFFERENCE IN LSM = -20.82, 95% CI 2-sided [-25.17 to -18.91], Standard Error of Mean 2.229
Statistical Analysis 2: Comparison: Maintenance Phase - CC-93538 360 mg Q2W vs Maintenance Phase - Placebo; Test type: Superiority; p < 0.0001, ANCOVA; DIFFERENCE IN LSM = -23.43, 95% CI 2-sided [-27.73 to -21.56], Standard Error of Mean 2.222

13. Secondary Outcome: Change From Baseline in Modified Daily Symptom Diary (mDSD) Composite Score at Week 24
Description: The mDSD composite score is evaluated over the prior 14-day period using the mDSD, which includes 6 primary questions. These questions assess solid food consumption that day (Q1), experience with trouble swallowing (Q2), food going down slowly (Q3), food getting stuck in the throat or chest (Q4), actions taken by participants to obtain relief (Q5), and any pain associated with swallowing (Q6). The daily symptom score (mDSD) is calculated by summing the responses to Q2, Q3, and Q4 (where "Yes" to any/all items equals 1, and "No" to all items equals 0), adding Q5 over the 14-day period prior to a visit, dividing by the number of measurable diary days over the 14-day period, and then multiplying by the length of the period (14). The daily symptom score ranges from 0 to 5, and the mDSD composite score ranges from 0 to 70 for the 14-day period. A higher composite diary score indicates more frequent and/or severe dysphagia symptoms.
Time Frame: Baseline (11 days prior to Day 1) and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo
Number analyzed (Participants) | 236 | 124
Score on a scale | -14.78 (11.353) | -10.93 (11.234)
Statistical Analysis 1: Comparison: Induction Phase - CC-93538 360 mg QW vs Induction Phase - Placebo; Test type: Superiority; p = 0.0005, ANCOVA; DIFFERENCE IN LSM = -4.10, 95% CI 2-sided [-6.40 to -1.80], Standard Error of Mean 1.174

14. Secondary Outcome: Change From Baseline in Modified Daily Symptom Diary (mDSD) Composite Score at Week 48
Description: as for outcome 13
Time Frame: Baseline (Day 1) , Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Maintenance Phase - CC-93538 360 mg QW | Maintenance Phase - CC-93538 360 mg Q2W | Maintenance Phase - Placebo
Number analyzed (Participants) | 100 | 101 | 75
score on a scale | -16.77 (11.297) | -16.45 (11.635) | -13.44 (10.862)
Statistical Analysis 1: Comparison: Maintenance Phase - CC-93538 360 mg QW vs Maintenance Phase - Placebo; Test type: Superiority; p = 0.0022, ANCOVA; DIFFERENCE IN LSM = -4.35, 95% CI 2-sided [-7.14 to -1.57], Standard Error of Mean 1.420
Statistical Analysis 2: Comparison: Maintenance Phase - CC-93538 360 mg QW vs Maintenance Phase - Placebo; Test type: Superiority; p = 0.0003, ANCOVA; Difference in LSM = -5.20, 95% CI 2-sided [-8.00 to -2.41], Standard Error of Mean 1.425

15. Secondary Outcome: Percentage of Participants With a ≥ 50% Decrease in Dysphagia Days(DD) From Baseline at Week 24
Description: Dysphagia Days (DD) was assessed using a modified daily symptom diary (mDSD). The DD was evaluated over the prior 14-day period using the mDSD, which includes 6 primary questions. These questions assess solid food consumption that day (Q1), experience with trouble swallowing (Q2), food going down slowly (Q3), food getting stuck in the throat or chest (Q4), actions taken by participants to obtain relief (Q5), and any pain associated with swallowing (Q6). The number of DD was normalized by calculating the number of diary days with a "yes" to any or all of Q2, Q3, and Q4 in the 14-day period prior to a visit, dividing by the number of measurable diary days in the 14-day period, and then multiplying by the length of the period (14). A measurable diary day for DD is defined as a diary day for which Questions 2 to 4 are answered. DD ranges from 0 to 14 for the 14-day period.
Time Frame: Baseline (11 days prior to Day 1) and Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo
Number analyzed (Participants) | 236 | 124
percentage of participants | 65.7 | 50.0
Statistical Analysis 1: Comparison: Induction Phase - CC-93538 360 mg QW vs Induction Phase - Placebo; Test type: Superiority; p = 0.0016, ANCOVA; DIFFERENCE IN RESPONSE RATE AFTER MI (%) = 16.9, 95% CI 2-sided [6.7 to 27.2]

16. Secondary Outcome: Percentage of Participants With a ≥ 50% Decrease in Dysphagia Days(DD) From Baseline at Week 48
Description: as for outcome 15
Time Frame: Baseline (11 days prior to Day 1) and Week 48
Population: The Intent-to-Treat (ITT)population consist of all randomized participants and analyzed according to their randomized treatment group regardless of whether or not the participant received IP CC-93538 or placebo. Number of participants with observed values at the specified timepoint are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance Phase - CC-93538 360 mg QW | Maintenance Phase - CC-93538 360 mg Q2W | Maintenance Phase - Placebo
Number analyzed (Participants) | 143 | 143 | 144
percentage of participants | 50.3 | 53.8 | 31.9

17. Secondary Outcome: Change From Baseline in Mean Dysphagia Days (DD) Through Week 24
Description: as for outcome 1
Time Frame: Baseline (Day 1), Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo
Number analyzed (Participants) | 264 | 144
days
  Week 2: number analyzed (Participants) | 262 | 139
  Week 2 | -1.26 (2.607) | -0.80 (2.651)
  Week 4: number analyzed (Participants) | 264 | 135
  Week 4 | -3.19 (4.073) | -1.75 (3.460)
  Week 8: number analyzed (Participants) | 255 | 132
  Week 8 | -5.04 (4.755) | -3.51 (4.132)
  Week 12: number analyzed (Participants) | 244 | 122
  Week 12 | -5.88 (5.071) | -3.88 (4.379)
  Week 16: number analyzed (Participants) | 235 | 121
  Week 16 | -6.39 (5.299) | -4.90 (4.851)
  Week 20: number analyzed (Participants) | 229 | 120
  Week 20 | -6.91 (5.321) | -4.98 (4.960)
  Week 24: number analyzed (Participants) | 236 | 124
  Week 24 | -6.85 (5.259) | -4.98 (5.075)

18. Secondary Outcome: Change From Baseline in Modified Daily Symptom Diary (mDSD) Composite Score Through Week 24
Description: as for outcome 13
Time Frame: Baseline (11 days prior to Day 1) and Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo
Number analyzed (Participants) | 264 | 139
Score on a scale
  Week 2: number analyzed (Participants) | 262 | 139
  Week 2 | -3.89 (7.126) | -3.25 (6.621)
  Week 4: number analyzed (Participants) | 264 | 135
  Week 4 | -8.02 (9.118) | -4.98 (8.902)
  Week 8: number analyzed (Participants) | 255 | 132
  Week 8 | -11.63 (10.515) | -7.59 (9.938)
  Week 12: number analyzed (Participants) | 244 | 122
  Week 12 | -13.22 (10.987) | -9.00 (10.051)
  Week 16: number analyzed (Participants) | 235 | 121
  Week 16 | -13.54 (11.623) | -10.43 (10.419)
  Week 20: number analyzed (Participants) | 229 | 120
  Week 20 | -14.71 (11.496) | -10.99 (10.353)
  Week 24: number analyzed (Participants) | 236 | 124
  Week 24 | -14.78 (11.353) | -10.93 (11.234)

19. Secondary Outcome: Time to First Event of Eosinophilic Esophagitis (EoE) Flare
Description: First incidence of corresponding EoE flare event for any participant was considered in the analysis. Median and 95% CI are from Kaplan-Meier estimates. Participants without an event of EoE flare or discontinued the study by the end of maintenance phase were censored, if they are a dropout, they are censored at study discontinuation date, otherwise they are censored at either last dose date or last visit, whichever was longer.
Time Frame: From first dose (Day 1) and Up to Week 48
Population: The Intent-to-Treat (ITT) population consist of all randomized participants and analyzed according to their randomized treatment group regardless of whether or not the participant received IP CC-93538 or placebo.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CC-93538 360 mg QW | CC-93538 360 mg QW/Q2W | Placebo
Number analyzed (Participants) | 143 | 143 | 144
days | NA [NA to NA] — Not Estimable due to inadequate number of events. | NA [NA to NA] — Not Estimable due to inadequate number of events. | NA [NA to NA] — Not Estimable due to inadequate number of events.

20. Secondary Outcome: Time to First Use of Rescue Medication
Description: First use of rescue therapy including EoE standard of care pharmacotherapy, dietary modification (e.g., food elimination diet), and/or dilation procedure. was considered in the analysis. Median and 95% CI are from Kaplan-Meier estimates. Participants without an event or discontinued the study by the end of maintenance phase were censored, if they are a dropout, they are censored at study discontinuation date, otherwise they are censored at either last dose date or last visit, whichever was longer.
Time Frame: From first dose (Day 1) and Up to Week 48
Population: The Intent-to-Treat (ITT)population consist of all randomized participants and analyzed according to their randomized treatment group regardless of whether or not the participant received IP CC-93538 or placebo.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CC-93538 360 mg QW | CC-93538 360 mg QW/Q2W | Placebo
Number analyzed (Participants) | 143 | 143 | 144
days | NA [NA to NA] — Not Estimable due to inadequate number of events. | NA [NA to NA] — Not Estimable due to inadequate number of events. | NA [NA to NA] — Not Estimable due to inadequate number of events.

21. Secondary Outcome: Percentage of Participants With Any Events of Use of Rescue Medication
Description: Use of rescue therapy including EoE standard of care pharmacotherapy, dietary modification (e.g., food elimination diet), and/or dilation procedure was considered in the analysis.
Time Frame: From first dose (Day 1) and up to Week 48
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | CC-93538 360 mg QW | CC-93538 360 mg QW/Q2W | Placebo
Number analyzed (Participants) | 143 | 143 | 144
percentage of participants | 4.9 | 7.0 | 13.9

22. Secondary Outcome: Percentage of Participants With Eosinophilic Esophagitis (EoE) Flare
Description: First incidence of corresponding EoE flare event for any participant was considered in the analysis.
Time Frame: From first dose (Day 1) and up to Week 48
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | CC-93538 360 mg QW | CC-93538 360 mg QW/Q2W | Placebo
Number analyzed (Participants) | 143 | 143 | 144
percentage of participants | 3.5 | 9.1 | 20.1

23. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From first dose (Day 1) till up to Week 48
Population: Safety population includes all the participants who received at least one dose of study treatment and analyzed based on the actual treatments they received.
Measure: Count of Participants; unit: Participants
Arm/Group | CC-93538 360 mg QW | CC-93538 360 mg QW/Q2W | Placebo
Number analyzed (Participants) | 167 | 117 | 143
Participants
  Treatment Emergent Adverse Events | 140 | 99 | 105
  Treatment Emergent Serious Adverse Events | 4 | 4 | 8
  Any Treatment Emergent Severe Adverse Events | 7 | 6 | 13
  Any Treatment Emergent Moderate Adverse Events | 68 | 55 | 48
  Any Treatment Emergent Mild Adverse Events | 65 | 38 | 44

24. Secondary Outcome: Number of Participants With Maximum Post-Baseline Clinical Laboratory Range Shift
Description: Blood samples were collected to assess clinical laboratory parameters. The row title contains parameter and category title contains shift. The category 'Normal to High' signifies the readings for the parameter were 'Normal' at baseline and it changed to 'High' post baseline.
Time Frame: From first dose (Day 1) till up to Week 48
Population: The Safety population consist of all randomized participants who received at least 1 dose of IP and analyzed based on the actual treatments they received.
Measure: Count of Participants; unit: Participants
Arm/Group | CC-93538 360 mg QW | CC-93538 360 mg QW/Q2W | Placebo
Number analyzed (Participants) | 167 | 117 | 143
Participants
  Sodium (mmol/L): Normal to Normal | 158 | 113 | 138
  Sodium (mmol/L): Normal to Low | 0 | 0 | 0
  Sodium (mmol/L): Normal to High | 7 | 4 | 4
  Sodium (mmol/L): Low to Normal | 0 | 0 | 1
  Sodium (mmol/L): Low to Low | 0 | 0 | 0
  Sodium (mmol/L): Low to High | 0 | 0 | 0
  Sodium (mmol/L): High to Normal | 1 | 0 | 0
  Sodium (mmol/L): High to Low | 0 | 0 | 0
  Sodium (mmol/L): High to High | 0 | 0 | 0
  Sodium (mmol/L): Missing | 1 | 0 | 0
  Potassium (mmol/L): Normal to Normal | 159 | 108 | 137
  Potassium (mmol/L): Normal to Low | 0 | 0 | 0
  Potassium (mmol/L): Normal to High | 6 | 9 | 6
  Potassium (mmol/L): Low to Normal | 1 | 0 | 0
  Potassium (mmol/L): Low to Low | 0 | 0 | 0
  Potassium (mmol/L): Low to High | 0 | 0 | 0
  Potassium (mmol/L): High to Normal | 0 | 0 | 0
  Potassium (mmol/L): High to Low | 0 | 0 | 0
  Potassium (mmol/L): High to High | 0 | 0 | 0
  Potassium (mmol/L): Missing | 1 | 0 | 0
  Chloride (mmol/L): Normal to Normal | 162 | 116 | 139
  Chloride (mmol/L): Normal to Low | 0 | 0 | 0
  Chloride (mmol/L): Normal to High | 3 | 1 | 3
  Chloride (mmol/L): Low to Normal | 1 | 0 | 1
  Chloride (mmol/L): Low to Low | 0 | 0 | 0
  Chloride (mmol/L): Low to High | 0 | 0 | 0
  Chloride (mmol/L): High to Normal | 0 | 0 | 0
  Chloride (mmol/L): High to Low | 0 | 0 | 0
  Chloride (mmol/L): High to High | 0 | 0 | 0
  Chloride (mmol/L): Missing | 1 | 0 | 0
  Calcium (mmol/L): Normal to Normal | 161 | 114 | 136
  Calcium (mmol/L): Normal to Low | 0 | 0 | 0
  Calcium (mmol/L): Normal to High | 2 | 3 | 3
  Calcium (mmol/L): Low to Normal | 2 | 0 | 1
  Calcium (mmol/L): Low to Low | 0 | 0 | 0
  Calcium (mmol/L): Low to High | 0 | 0 | 0
  Calcium (mmol/L): High to Normal | 1 | 0 | 3
  Calcium (mmol/L): High to Low | 0 | 0 | 0
  Calcium (mmol/L): High to High | 0 | 0 | 0
  Calcium (mmol/L): Missing | 1 | 0 | 0
  Magnesium (mmol/L): Normal to Normal | 162 | 111 | 138
  Magnesium (mmol/L): Normal to Low | 0 | 0 | 0
  Magnesium (mmol/L): Normal to High | 3 | 4 | 4
  Magnesium (mmol/L): Low to Normal | 0 | 0 | 0
  Magnesium (mmol/L): Low to Low | 0 | 0 | 0
  Magnesium (mmol/L): Low to High | 0 | 0 | 0
  Magnesium (mmol/L): High to Normal | 0 | 1 | 0
  Magnesium (mmol/L): High to Low | 0 | 0 | 0
  Magnesium (mmol/L): High to High | 1 | 1 | 1
  Magnesium (mmol/L): Missing | 1 | 0 | 0
  Phosphate (mmol/L): Normal to Normal | 159 | 112 | 136
  Phosphate (mmol/L): Normal to Low | 0 | 0 | 0
  Phosphate (mmol/L): Normal to High | 4 | 4 | 5
  Phosphate (mmol/L): Low to Normal | 2 | 0 | 1
  Phosphate (mmol/L): Low to Low | 0 | 0 | 0
  Phosphate (mmol/L): Low to High | 0 | 0 | 0
  Phosphate (mmol/L): High to Normal | 0 | 0 | 1
  Phosphate (mmol/L): High to Low | 0 | 0 | 0
  Phosphate (mmol/L): High to High | 1 | 1 | 0
  Phosphate (mmol/L): Missing | 1 | 0 | 0
  Blood Urea Nitrogen (mmol/L): Normal to Normal | 160 | 108 | 137
  Blood Urea Nitrogen (mmol/L): Normal to Low | 0 | 0 | 0
  Blood Urea Nitrogen (mmol/L): Normal to High | 6 | 8 | 6
  Blood Urea Nitrogen (mmol/L): Low to Normal | 0 | 0 | 0
  Blood Urea Nitrogen (mmol/L): Low to Low | 0 | 0 | 0
  Blood Urea Nitrogen (mmol/L): Low to High | 0 | 0 | 0
  Blood Urea Nitrogen (mmol/L): High to Normal | 0 | 0 | 0
  Blood Urea Nitrogen (mmol/L): High to Low | 0 | 0 | 0
  Blood Urea Nitrogen (mmol/L): High to High | 0 | 1 | 0
  Blood Urea Nitrogen (mmol/L): Missing | 1 | 0 | 0
  Glucose (mmol/L): Normal to Normal | 101 | 69 | 88
  Glucose (mmol/L): Normal to Low | 0 | 0 | 0
  Glucose (mmol/L): Normal to High | 40 | 36 | 30
  Glucose (mmol/L): Low to Normal | 3 | 0 | 2
  Glucose (mmol/L): Low to Low | 0 | 0 | 0
  Glucose (mmol/L): Low to High | 0 | 0 | 0
  Glucose (mmol/L): High to Normal | 5 | 2 | 2
  Glucose (mmol/L): High to Low | 0 | 0 | 0
  Glucose (mmol/L): High to High | 17 | 10 | 21
  Glucose (mmol/L): Missing | 1 | 0 | 0
  Albumin (g/L): Normal to Normal | 94 | 60 | 76
  Albumin (g/L): Normal to Low | 0 | 0 | 0
  Albumin (g/L): Normal to High | 37 | 30 | 35
  Albumin (g/L): Low to Normal | 0 | 0 | 0
  Albumin (g/L): Low to Low | 0 | 0 | 0
  Albumin (g/L): Low to High | 0 | 0 | 0
  Albumin (g/L): High to Normal | 10 | 2 | 9
  Albumin (g/L): High to Low | 0 | 0 | 0
  Albumin (g/L): High to High | 25 | 25 | 23
  Albumin (g/L): Missing | 1 | 0 | 0
  Alkaline Phosphatase (U/L): Normal to Normal | 140 | 104 | 129
  Alkaline Phosphatase (U/L): Normal to Low | 0 | 0 | 0
  Alkaline Phosphatase (U/L): Normal to High | 9 | 4 | 7
  Alkaline Phosphatase (U/L): Low to Normal | 1 | 2 | 1
  Alkaline Phosphatase (U/L): Low to Low | 1 | 0 | 0
  Alkaline Phosphatase (U/L): Low to High | 0 | 0 | 0
  Alkaline Phosphatase (U/L): High to Normal | 3 | 1 | 1
  Alkaline Phosphatase (U/L): High to Low | 0 | 0 | 0
  Alkaline Phosphatase (U/L): High to High | 12 | 6 | 5
  Alkaline Phosphatase (U/L): Missing | 1 | 0 | 0
  Creatinine (umol/L): Normal to Normal | 152 | 107 | 131
  Creatinine (umol/L): Normal to Low | 0 | 0 | 0
  Creatinine (umol/L): Normal to High | 7 | 6 | 7
  Creatinine (umol/L): Low to Normal | 1 | 0 | 0
  Creatinine (umol/L): Low to Low | 0 | 0 | 0
  Creatinine (umol/L): Low to High | 0 | 0 | 0
  Creatinine (umol/L): High to Normal | 1 | 0 | 1
  Creatinine (umol/L): High to Low | 0 | 0 | 0
  Creatinine (umol/L): High to High | 5 | 4 | 4
  Creatinine (umol/L): Missing | 1 | 0 | 0
  Creatine Kinase (U/L): Normal to Normal | 115 | 64 | 100
  Creatine Kinase (U/L): Normal to Low | 0 | 0 | 0
  Creatine Kinase (U/L): Normal to High | 39 | 39 | 36
  Creatine Kinase (U/L): Low to Normal | 1 | 0 | 0
  Creatine Kinase (U/L): Low to Low | 0 | 0 | 0
  Creatine Kinase (U/L): Low to High | 0 | 0 | 0
  Creatine Kinase (U/L): High to Normal | 4 | 4 | 0
  Creatine Kinase (U/L): High to Low | 0 | 0 | 0
  Creatine Kinase (U/L): High to High | 7 | 10 | 7
  Creatine Kinase (U/L): Missing | 1 | 0 | 0
  Alanine Aminotransferase (U/L): Normal to Normal | 131 | 88 | 111
  Alanine Aminotransferase (U/L): Normal to Low | 0 | 0 | 0
  Alanine Aminotransferase (U/L): Normal to High | 22 | 22 | 22
  Alanine Aminotransferase (U/L): Low to Normal | 0 | 0 | 0
  Alanine Aminotransferase (U/L): Low to Low | 0 | 0 | 0
  Alanine Aminotransferase (U/L): Low to High | 0 | 0 | 0
  Alanine Aminotransferase (U/L): High to Normal | 2 | 1 | 3
  Alanine Aminotransferase (U/L): High to Low | 0 | 0 | 0
  Alanine Aminotransferase (U/L): High to High | 11 | 6 | 7
  Alanine Aminotransferase (U/L): Missing | 1 | 0 | 0
  Aspartate Aminotransferase (U/L): Normal to Normal | 143 | 93 | 120
  Aspartate Aminotransferase (U/L): Normal to Low | 0 | 0 | 0
  Aspartate Aminotransferase (U/L): Normal to High | 18 | 20 | 17
  Aspartate Aminotransferase (U/L): Low to Normal | 0 | 0 | 1
  Aspartate Aminotransferase (U/L): Low to Low | 0 | 0 | 0
  Aspartate Aminotransferase (U/L): Low to High | 0 | 0 | 0
  Aspartate Aminotransferase (U/L): High to Normal | 2 | 0 | 1
  Aspartate Aminotransferase (U/L): High to Low | 0 | 0 | 0
  Aspartate Aminotransferase (U/L): High to High | 3 | 4 | 4
  Aspartate Aminotransferase (U/L): Missing | 1 | 0 | 0
  Gamma Glutamyl Transferase (U/L): Normal to Normal | 149 | 103 | 122
  Gamma Glutamyl Transferase (U/L): Normal to Low | 0 | 0 | 0
  Gamma Glutamyl Transferase (U/L): Normal to High | 5 | 8 | 9
  Gamma Glutamyl Transferase (U/L): Low to Normal | 0 | 1 | 1
  Gamma Glutamyl Transferase (U/L): Low to Low | 2 | 0 | 0
  Gamma Glutamyl Transferase (U/L): Low to High | 0 | 0 | 0
  Gamma Glutamyl Transferase (U/L): High to Normal | 2 | 0 | 1
  Gamma Glutamyl Transferase (U/L): High to Low | 0 | 0 | 0
  Gamma Glutamyl Transferase (U/L): High to High | 8 | 5 | 10
  Gamma Glutamyl Transferase (U/L): Missing | 1 | 0 | 0
  Amylase (U/L): Normal to Normal | 128 | 98 | 127
  Amylase (U/L): Normal to Low | 1 | 0 | 0
  Amylase (U/L): Normal to High | 15 | 9 | 4
  Amylase (U/L): Low to Normal | 4 | 2 | 4
  Amylase (U/L): Low to Low | 3 | 0 | 0
  Amylase (U/L): Low to High | 0 | 0 | 0
  Amylase (U/L): High to Normal | 3 | 0 | 0
  Amylase (U/L): High to Low | 0 | 0 | 0
  Amylase (U/L): High to High | 12 | 8 | 8
  Amylase (U/L): Missing | 1 | 0 | 0
  Total Bilirubin (umol/L): Normal to Normal | 146 | 106 | 123
  Total Bilirubin (umol/L): Normal to Low | 1 | 0 | 0
  Total Bilirubin (umol/L): Normal to High | 8 | 5 | 9
  Total Bilirubin (umol/L): Low to Normal | 5 | 2 | 6
  Total Bilirubin (umol/L): Low to Low | 0 | 0 | 0
  Total Bilirubin (umol/L): Low to High | 0 | 0 | 0
  Total Bilirubin (umol/L): High to Normal | 2 | 0 | 0
  Total Bilirubin (umol/L): High to Low | 0 | 0 | 0
  Total Bilirubin (umol/L): High to High | 4 | 4 | 5
  Total Bilirubin (umol/L): Missing | 1 | 0 | 0
  Direct Bilirubin (umol/L): Normal to Normal | 165 | 117 | 143
  Direct Bilirubin (umol/L): Normal to Low | 0 | 0 | 0
  Direct Bilirubin (umol/L): Normal to High | 1 | 0 | 0
  Direct Bilirubin (umol/L): Low to Normal | 0 | 0 | 0
  Direct Bilirubin (umol/L): Low to Low | 0 | 0 | 0
  Direct Bilirubin (umol/L): Low to High | 0 | 0 | 0
  Direct Bilirubin (umol/L): High to Normal | 0 | 0 | 0
  Direct Bilirubin (umol/L): High to Low | 0 | 0 | 0
  Direct Bilirubin (umol/L): High to High | 0 | 0 | 0
  Direct Bilirubin (umol/L): Missing | 1 | 0 | 0
  C Reactive Protein (mg/L): Normal to Normal | 107 | 70 | 85
  C Reactive Protein (mg/L): Normal to Low | 0 | 0 | 0
  C Reactive Protein (mg/L): Normal to High | 34 | 25 | 35
  C Reactive Protein (mg/L): Low to Normal | 0 | 0 | 0
  C Reactive Protein (mg/L): Low to Low | 0 | 0 | 0
  C Reactive Protein (mg/L): Low to High | 0 | 0 | 0
  C Reactive Protein (mg/L): High to Normal | 1 | 4 | 4
  C Reactive Protein (mg/L): High to Low | 0 | 0 | 0
  C Reactive Protein (mg/L): High to High | 18 | 9 | 13
  C Reactive Protein (mg/L): Missing | 7 | 9 | 6
  Cholesterol (mmol/L): Normal to Normal | 116 | 91 | 102
  Cholesterol (mmol/L): Normal to Low | 3 | 3 | 1
  Cholesterol (mmol/L): Normal to High | 5 | 4 | 5
  Cholesterol (mmol/L): Low to Normal | 14 | 5 | 6
  Cholesterol (mmol/L): Low to Low | 2 | 5 | 9
  Cholesterol (mmol/L): Low to High | 0 | 0 | 0
  Cholesterol (mmol/L): High to Normal | 3 | 3 | 2
  Cholesterol (mmol/L): High to Low | 0 | 0 | 0
  Cholesterol (mmol/L): High to High | 1 | 3 | 2
  Cholesterol (mmol/L): Missing | 23 | 3 | 16
  Triglycerides (mmol/L): Normal to Normal | 124 | 93 | 105
  Triglycerides (mmol/L): Normal to Low | 0 | 1 | 2
  Triglycerides (mmol/L): Normal to High | 7 | 3 | 4
  Triglycerides (mmol/L): Low to Normal | 3 | 6 | 3
  Triglycerides (mmol/L): Low to Low | 0 | 1 | 0
  Triglycerides (mmol/L): Low to High | 0 | 0 | 0
  Triglycerides (mmol/L): High to Normal | 6 | 3 | 7
  Triglycerides (mmol/L): High to Low | 0 | 0 | 0
  Triglycerides (mmol/L): High to High | 3 | 6 | 5
  Triglycerides (mmol/L): Missing | 24 | 4 | 17
  HDL Cholesterol (mmol/L): Normal to Normal | 63 | 37 | 65
  HDL Cholesterol (mmol/L): Normal to Low | 5 | 1 | 3
  HDL Cholesterol (mmol/L): Normal to High | 15 | 10 | 9
  HDL Cholesterol (mmol/L): Low to Normal | 4 | 14 | 11
  HDL Cholesterol (mmol/L): Low to Low | 18 | 22 | 14
  HDL Cholesterol (mmol/L): Low to High | 0 | 0 | 0
  HDL Cholesterol (mmol/L): High to Normal | 5 | 5 | 5
  HDL Cholesterol (mmol/L): High to Low | 0 | 0 | 0
  HDL Cholesterol (mmol/L): High to High | 33 | 25 | 19
  HDL Cholesterol (mmol/L): Missing | 24 | 3 | 17
  LDL Cholesterol (mmol/L): Normal to Normal | 111 | 88 | 101
  LDL Cholesterol (mmol/L): Normal to Low | 2 | 3 | 3
  LDL Cholesterol (mmol/L): Normal to High | 5 | 4 | 5
  LDL Cholesterol (mmol/L): Low to Normal | 12 | 9 | 3
  LDL Cholesterol (mmol/L): Low to Low | 8 | 4 | 10
  LDL Cholesterol (mmol/L): Low to High | 0 | 0 | 0
  LDL Cholesterol (mmol/L): High to Normal | 2 | 0 | 2
  LDL Cholesterol (mmol/L): High to Low | 0 | 0 | 0
  LDL Cholesterol (mmol/L): High to High | 2 | 2 | 1
  LDL Cholesterol (mmol/L): Missing | 25 | 7 | 18
  Erythrocytes (10^12/L): Normal to Normal | 154 | 113 | 137
  Erythrocytes (10^12/L): Normal to Low | 1 | 0 | 0
  Erythrocytes (10^12/L): Normal to High | 2 | 0 | 0
  Erythrocytes (10^12/L): Low to Normal | 5 | 2 | 3
  Erythrocytes (10^12/L): Low to Low | 1 | 1 | 1
  Erythrocytes (10^12/L): Low to High | 0 | 0 | 0
  Erythrocytes (10^12/L): High to Normal | 0 | 0 | 0
  Erythrocytes (10^12/L): High to Low | 0 | 0 | 0
  Erythrocytes (10^12/L): High to High | 1 | 1 | 2
  Erythrocytes (10^12/L): Missing | 3 | 0 | 0
  Leukocytes (10^9/L): Normal to Normal | 144 | 96 | 125
  Leukocytes (10^9/L): Normal to Low | 2 | 0 | 0
  Leukocytes (10^9/L): Normal to High | 9 | 11 | 7
  Leukocytes (10^9/L): Low to Normal | 4 | 7 | 6
  Leukocytes (10^9/L): Low to Low | 0 | 0 | 0
  Leukocytes (10^9/L): Low to High | 0 | 0 | 0
  Leukocytes (10^9/L): High to Normal | 2 | 1 | 3
  Leukocytes (10^9/L): High to Low | 0 | 0 | 0
  Leukocytes (10^9/L): High to High | 3 | 2 | 2
  Leukocytes (10^9/L): Missing | 3 | 0 | 0
  Basophils (10^9/L): Normal to Normal | 159 | 112 | 141
  Basophils (10^9/L): Normal to Low | 0 | 0 | 0
  Basophils (10^9/L): Normal to High | 5 | 5 | 2
  Basophils (10^9/L): Low to Normal | 0 | 0 | 0
  Basophils (10^9/L): Low to Low | 0 | 0 | 0
  Basophils (10^9/L): Low to High | 0 | 0 | 0
  Basophils (10^9/L): High to Normal | 0 | 0 | 0
  Basophils (10^9/L): High to Low | 0 | 0 | 0
  Basophils (10^9/L): High to High | 0 | 0 | 0
  Basophils (10^9/L): Missing | 3 | 0 | 0
  Basophils/Leukocytes (%): Normal to Normal | 124 | 75 | 113
  Basophils/Leukocytes (%): Normal to Low | 0 | 0 | 0
  Basophils/Leukocytes (%): Normal to High | 36 | 37 | 26
  Basophils/Leukocytes (%): Low to Normal | 0 | 0 | 0
  Basophils/Leukocytes (%): Low to Low | 0 | 0 | 0
  Basophils/Leukocytes (%): Low to High | 0 | 0 | 0
  Basophils/Leukocytes (%): High to Normal | 2 | 3 | 4
  Basophils/Leukocytes (%): High to Low | 0 | 0 | 0
  Basophils/Leukocytes (%): High to High | 2 | 2 | 0
  Basophils/Leukocytes (%): Missing | 3 | 0 | 0
  Eosinophils (10^9/L): Normal to Normal | 115 | 81 | 89
  Eosinophils (10^9/L): Normal to Low | 0 | 0 | 0
  Eosinophils (10^9/L): Normal to High | 32 | 22 | 41
  Eosinophils (10^9/L): Low to Normal | 0 | 0 | 0
  Eosinophils (10^9/L): Low to Low | 0 | 0 | 0
  Eosinophils (10^9/L): Low to High | 0 | 0 | 0
  Eosinophils (10^9/L): High to Normal | 3 | 1 | 3
  Eosinophils (10^9/L): High to Low | 0 | 0 | 0
  Eosinophils (10^9/L): High to High | 14 | 13 | 10
  Eosinophils (10^9/L): Missing | 3 | 0 | 0
  Eosinophils/Leukocytes (%): Normal to Normal | 88 | 56 | 54
  Eosinophils/Leukocytes (%): Normal to Low | 0 | 0 | 0
  Eosinophils/Leukocytes (%): Normal to High | 39 | 26 | 45
  Eosinophils/Leukocytes (%): Low to Normal | 0 | 0 | 0
  Eosinophils/Leukocytes (%): Low to Low | 0 | 0 | 0
  Eosinophils/Leukocytes (%): Low to High | 0 | 0 | 0
  Eosinophils/Leukocytes (%): High to Normal | 7 | 7 | 4
  Eosinophils/Leukocytes (%): High to Low | 0 | 0 | 0
  Eosinophils/Leukocytes (%): High to High | 30 | 28 | 40
  Eosinophils/Leukocytes (%): Missing | 3 | 0 | 0
  Lymphocytes (10^9/L): Normal to Normal | 157 | 113 | 138
  Lymphocytes (10^9/L): Normal to Low | 0 | 0 | 0
  Lymphocytes (10^9/L): Normal to High | 6 | 1 | 4
  Lymphocytes (10^9/L): Low to Normal | 1 | 3 | 1
  Lymphocytes (10^9/L): Low to Low | 0 | 0 | 0
  Lymphocytes (10^9/L): Low to High | 0 | 0 | 0
  Lymphocytes (10^9/L): High to Normal | 0 | 0 | 0
  Lymphocytes (10^9/L): High to Low | 0 | 0 | 0
  Lymphocytes (10^9/L): High to High | 0 | 0 | 0
  Lymphocytes (10^9/L): Missing | 3 | 0 | 0
  Lymphocytes/Leukocytes (%): Normal to Normal | 148 | 108 | 131
  Lymphocytes/Leukocytes (%): Normal to Low | 0 | 0 | 0
  Lymphocytes/Leukocytes (%): Normal to High | 14 | 6 | 8
  Lymphocytes/Leukocytes (%): Low to Normal | 1 | 1 | 3
  Lymphocytes/Leukocytes (%): Low to Low | 0 | 0 | 0
  Lymphocytes/Leukocytes (%): Low to High | 0 | 0 | 0
  Lymphocytes/Leukocytes (%): High to Normal | 0 | 0 | 1
  Lymphocytes/Leukocytes (%): High to Low | 0 | 0 | 0
  Lymphocytes/Leukocytes (%): High to High | 1 | 2 | 0
  Lymphocytes/Leukocytes (%): Missing | 3 | 0 | 0
  Monocytes (10^9/L): Normal to Normal | 154 | 109 | 134
  Monocytes (10^9/L): Normal to Low | 0 | 0 | 0
  Monocytes (10^9/L): Normal to High | 2 | 0 | 1
  Monocytes (10^9/L): Low to Normal | 5 | 7 | 3
  Monocytes (10^9/L): Low to Low | 2 | 1 | 4
  Monocytes (10^9/L): Low to High | 0 | 0 | 0
  Monocytes (10^9/L): High to Normal | 0 | 0 | 0
  Monocytes (10^9/L): High to Low | 0 | 0 | 0
  Monocytes (10^9/L): High to High | 1 | 0 | 1
  Monocytes (10^9/L): Missing | 3 | 0 | 0
  Monocytes/Leukocytes (%): Normal to Normal | 140 | 97 | 124
  Monocytes/Leukocytes (%): Normal to Low | 0 | 0 | 0
  Monocytes/Leukocytes (%): Normal to High | 18 | 14 | 14
  Monocytes/Leukocytes (%): Low to Normal | 2 | 1 | 3
  Monocytes/Leukocytes (%): Low to Low | 0 | 0 | 0
  Monocytes/Leukocytes (%): Low to High | 0 | 0 | 0
  Monocytes/Leukocytes (%): High to Normal | 0 | 0 | 1
  Monocytes/Leukocytes (%): High to Low | 0 | 0 | 0
  Monocytes/Leukocytes (%): High to High | 4 | 5 | 1
  Monocytes/Leukocytes (%): Missing | 3 | 0 | 0
  NEUTROPHILS, SEGMENTED (10^9/L): Normal to Normal | 138 | 93 | 120
  NEUTROPHILS, SEGMENTED (10^9/L): Normal to Low | 3 | 0 | 0
  NEUTROPHILS, SEGMENTED (10^9/L): Normal to High | 12 | 10 | 12
  NEUTROPHILS, SEGMENTED (10^9/L): Low to Normal | 7 | 10 | 5
  NEUTROPHILS, SEGMENTED (10^9/L): Low to Low | 0 | 0 | 0
  NEUTROPHILS, SEGMENTED (10^9/L): Low to High | 0 | 0 | 1
  NEUTROPHILS, SEGMENTED (10^9/L): High to Normal | 1 | 1 | 3
  NEUTROPHILS, SEGMENTED (10^9/L): High to Low | 0 | 0 | 0
  NEUTROPHILS, SEGMENTED (10^9/L): High to High | 3 | 3 | 2
  NEUTROPHILS, SEGMENTED (10^9/L): Missing | 3 | 0 | 0
  NEUTROPHILS/LEUKOCYTES (%): Normal to Normal | 142 | 101 | 122
  NEUTROPHILS/LEUKOCYTES (%): Normal to Low | 1 | 0 | 0
  NEUTROPHILS/LEUKOCYTES (%): Normal to High | 15 | 7 | 14
  NEUTROPHILS/LEUKOCYTES (%): Low to Normal | 4 | 7 | 3
  NEUTROPHILS/LEUKOCYTES (%): Low to Low | 0 | 0 | 0
  NEUTROPHILS/LEUKOCYTES (%): Low to High | 0 | 0 | 0
  NEUTROPHILS/LEUKOCYTES (%): High to Normal | 1 | 1 | 3
  NEUTROPHILS/LEUKOCYTES (%): High to Low | 0 | 0 | 0
  NEUTROPHILS/LEUKOCYTES (%): High to High | 1 | 1 | 1
  NEUTROPHILS/LEUKOCYTES (%): Missing | 3 | 0 | 0
  PLATELETS (10^9/L): Normal to Normal | 153 | 102 | 128
  PLATELETS (10^9/L): Normal to Low | 0 | 0 | 0
  PLATELETS (10^9/L): Normal to High | 7 | 11 | 11
  PLATELETS (10^9/L): Low to Normal | 1 | 1 | 2
  PLATELETS (10^9/L): Low to Low | 0 | 0 | 0
  PLATELETS (10^9/L): Low to High | 0 | 0 | 0
  PLATELETS (10^9/L): High to Normal | 1 | 0 | 0
  PLATELETS (10^9/L): High to Low | 0 | 0 | 0
  PLATELETS (10^9/L): High to High | 1 | 3 | 2
  PLATELETS (10^9/L): Missing | 4 | 0 | 0
  HEMOGLOBIN (g/L): Normal to Normal | 158 | 115 | 142
  HEMOGLOBIN (g/L): Normal to Low | 1 | 0 | 0
  HEMOGLOBIN (g/L): Normal to High | 4 | 0 | 0
  HEMOGLOBIN (g/L): Low to Normal | 1 | 0 | 1
  HEMOGLOBIN (g/L): Low to Low | 0 | 1 | 0
  HEMOGLOBIN (g/L): Low to High | 0 | 0 | 0
  HEMOGLOBIN (g/L): High to Normal | 0 | 0 | 0
  HEMOGLOBIN (g/L): High to Low | 0 | 0 | 0
  HEMOGLOBIN (g/L): High to High | 0 | 1 | 0
  HEMOGLOBIN (g/L): Missing | 3 | 0 | 0
  HEMATOCRIT (VOLUME FRACTION): Normal to Normal | 158 | 110 | 140
  HEMATOCRIT (VOLUME FRACTION): Normal to Low | 1 | 0 | 0
  HEMATOCRIT (VOLUME FRACTION): Normal to High | 4 | 2 | 0
  HEMATOCRIT (VOLUME FRACTION): Low to Normal | 1 | 4 | 2
  HEMATOCRIT (VOLUME FRACTION): Low to Low | 0 | 0 | 0
  HEMATOCRIT (VOLUME FRACTION): Low to High | 0 | 0 | 0
  HEMATOCRIT (VOLUME FRACTION): High to Normal | 0 | 0 | 0
  HEMATOCRIT (VOLUME FRACTION): High to Low | 0 | 0 | 0
  HEMATOCRIT (VOLUME FRACTION): High to High | 0 | 1 | 0
  HEMATOCRIT (VOLUME FRACTION): Missing | 3 | 0 | 1
  ERYTHROCYTES MEAN CORPUSCULAR VOLUME (Femtoliter): Normal to Normal | 128 | 90 | 120
  ERYTHROCYTES MEAN CORPUSCULAR VOLUME (Femtoliter): Normal to Low | 0 | 0 | 0
  ERYTHROCYTES MEAN CORPUSCULAR VOLUME (Femtoliter): Normal to High | 24 | 16 | 14
  ERYTHROCYTES MEAN CORPUSCULAR VOLUME (Femtoliter): Low to Normal | 6 | 3 | 4
  ERYTHROCYTES MEAN CORPUSCULAR VOLUME (Femtoliter): Low to Low | 1 | 2 | 1
  ERYTHROCYTES MEAN CORPUSCULAR VOLUME (Femtoliter): Low to High | 0 | 0 | 0
  ERYTHROCYTES MEAN CORPUSCULAR VOLUME (Femtoliter): High to Normal | 1 | 1 | 0
  ERYTHROCYTES MEAN CORPUSCULAR VOLUME (Femtoliter): High to Low | 0 | 0 | 0
  ERYTHROCYTES MEAN CORPUSCULAR VOLUME (Femtoliter): High to High | 4 | 5 | 3
  ERYTHROCYTES MEAN CORPUSCULAR VOLUME (Femtoliter): Missing | 3 | 0 | 1
  ERYTHROCTES MEAN CORPUSCULAR HEMOGLOBIN (picogram): Normal to Normal | 160 | 115 | 141
  ERYTHROCTES MEAN CORPUSCULAR HEMOGLOBIN (picogram): Normal to Low | 0 | 0 | 0
  ERYTHROCTES MEAN CORPUSCULAR HEMOGLOBIN (picogram): Normal to High | 0 | 0 | 0
  ERYTHROCTES MEAN CORPUSCULAR HEMOGLOBIN (picogram): Low to Normal | 3 | 0 | 1
  ERYTHROCTES MEAN CORPUSCULAR HEMOGLOBIN (picogram): Low to Low | 1 | 2 | 1
  ERYTHROCTES MEAN CORPUSCULAR HEMOGLOBIN (picogram): Low to High | 0 | 0 | 0
  ERYTHROCTES MEAN CORPUSCULAR HEMOGLOBIN (picogram): High to Normal | 0 | 0 | 0
  ERYTHROCTES MEAN CORPUSCULAR HEMOGLOBIN (picogram): High to Low | 0 | 0 | 0
  ERYTHROCTES MEAN CORPUSCULAR HEMOGLOBIN (picogram): High to High | 0 | 0 | 0
  ERYTHROCTES MEAN CORPUSCULAR HEMOGLOBIN (picogram): Missing | 3 | 0 | 0
  ERY. MEAN CORPUSCULAR HGB CONCENTRATION (g/L): Normal to Normal | 164 | 114 | 140
  ERY. MEAN CORPUSCULAR HGB CONCENTRATION (g/L): Normal to Low | 0 | 0 | 0
  ERY. MEAN CORPUSCULAR HGB CONCENTRATION (g/L): Normal to High | 0 | 0 | 0
  ERY. MEAN CORPUSCULAR HGB CONCENTRATION (g/L): Low to Normal | 0 | 3 | 2
  ERY. MEAN CORPUSCULAR HGB CONCENTRATION (g/L): Low to Low | 0 | 0 | 0
  ERY. MEAN CORPUSCULAR HGB CONCENTRATION (g/L): Low to High | 0 | 0 | 0
  ERY. MEAN CORPUSCULAR HGB CONCENTRATION (g/L): High to Normal | 0 | 0 | 0
  ERY. MEAN CORPUSCULAR HGB CONCENTRATION (g/L): High to Low | 0 | 0 | 0
  ERY. MEAN CORPUSCULAR HGB CONCENTRATION (g/L): High to High | 0 | 0 | 0
  ERY. MEAN CORPUSCULAR HGB CONCENTRATION (g/L): Missing | 3 | 0 | 1

25. Secondary Outcome: Number of Participants With Post-Baseline Vital Sign Abnormalities
Description: Vital signs like feart rate (beats per minute) and systolic blood pressure (mmHg) and diastolic blood pressure (mmHg) was measured to assess the abnormalities.
Time Frame: From first dose (Day 1) till up to Week 48
Population: The Safety population consist of all randomized participants who received at least 1 dose of IP and analyzed based on the actual treatments they received. Only number of participants with observed values at specified timepoints are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CC-93538 360 mg QW | CC-93538 360 mg QW/Q2W | Placebo
Number analyzed (Participants) | 167 | 117 | 143
Participants
  Hear rate (> 100 AND CHANGE FROM BASELINE > 30) | 6 | 1 | 3
  Hear rate (< 55 AND CHANGE FROM BASELINE < -15) | 0 | 0 | 0
  SBP (> 140 AND CHANGE FROM BASELINE > 20) | 16 | 11 | 15
  SBP (< 90 AND CHANGE FROM BASELINE < -20) | 0 | 0 | 0
  DBP > 90 AND CHANGE FROM BASELINE > 10 | 18 | 21 | 25
  DBP < 55 AND CHANGE FROM BASELINE < -10 | 4 | 6 | 8

26. Secondary Outcome: Change From Baseline in Physical Parameters - Height at Week 24
Description: Height was measured at specified timepoints to assess the change from baseline.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo
Number analyzed (Participants) | 225 | 115
cm | 0.30 (1.479) | -0.08 (0.932)

27. Secondary Outcome: Change From Baseline in Physical Parameters - Height at Week 48
Description: Height was measured at specified timepoints to assess the change from baseline.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maintenance Phase - CC-93538 360 mg QW | Maintenance Phase - CC-93538 360 mg Q2W | Maintenance Phase - Placebo
Number analyzed (Participants) | 88 | 96 | 75
cm | 0.42 (1.929) | 0.42 (1.973) | 0.12 (1.114)

28. Secondary Outcome: Change From Baseline in Physical Parameters - Weight at Week 24
Description: Weight was measured at specified timepoints to assess the change from baseline.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo
Number analyzed (Participants) | 257 | 133
kg | 0.35 (3.369) | 0.24 (3.108)

29. Secondary Outcome: Change From Baseline in Physical Parameters - Weight at Week 48
Description: Weight was measured at specified timepoints to assess the change from baseline.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Maintenance Phase - CC-93538 360 mg QW | Maintenance Phase - CC-93538 360 mg Q2W | Maintenance Phase - Placebo
Number analyzed (Participants) | 107 | 110 | 82
cm | 0.11 (4.908) | 1.26 (4.766) | 0.22 (4.270)

30. Secondary Outcome: Change From Baseline in Physical Parameters - Body Mass Index at Week 24
Description: Data was collected for height and weight to assess body mass index.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Induction Phase - CC-93538 360 mg QW | Induction Phase - Placebo
Number analyzed (Participants) | 256 | 133
kg/m^2 | 0.044 (1.1629) | 0.084 (1.0676)

31. Secondary Outcome: Change From Baseline in Physical Parameters - Body Mass Index at Week 48
Description: Data was collected for height and weight to assess body mass index.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Maintenance Phase - CC-93538 360 mg QW | Maintenance Phase - CC-93538 360 mg Q2W | Maintenance Phase - Placebo
Number analyzed (Participants) | 106 | 110 | 82
kg/m^2 | -0.074 (1.6716) | 0.350 (1.5218) | 0.037 (1.4223)

32. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA)
Description: ADA status were categorized as Baseline ADA Positive: Pre-existing Immunoreactivity (baseline positive and 1) post baseline negative or 2) titer < 4-fold baseline titer). NAb+/baseline ADA+: At least one ADA positive sample with positive NAb in participant with pre-existing immunoreactivity. ADA Positive Status: 1) at least one positive response post first dose given negative or missing baseline; or 2) at least one post-baseline with titer greater than or equal to 4-fold of baseline titer given positive baseline. NAb+/ADA+: At least one ADA positive sample with positive NAb in ADA positive participant.
Time Frame: Pre-dose Week 24 and Pre-dose Week 48
Population: The Pharmacokinetic population consist of all randomized participants who received at least one dose of CC-93538 and have any available concentration data.
Measure: Count of Participants; unit: Participants
Arm/Group | CC-93538 360 mg QW | CC-93538 360 mg QW/Q2W
Number analyzed (Participants) | 167 | 117
Participants
  BASELINE ADA POSITIVE (Week 24) | 6 | 5
  BASELINE ADA POSITIVE (Week 48) | 4 | 6
  NAB+/BASELINE ADA+ (Week 24) | 2 | 1
  NAB+/BASELINE ADA+ (Week 48) | 1 | 1
  ADA POSITIVE (Week 24) | 12 | 13
  ADA POSITIVE (Week 48) | 8 | 12
  NAB+/ADA+ (Week 24) | 4 | 7
  NAB+/ADA+ (Week 48) | 1 | 7

33. Secondary Outcome: Serum Trough Concentration of CC-93538 at Week 24 and Week 48
Description: Blood samples were collected to assess trough concentration of CC-93538. The Evaluable PK population is defined as all participants in the PK population who have at least one evaluable trough concentration.
Time Frame: Pre-dose Week 24 and Pre-dose Week 48
Population: The PK population will consist of all randomized participants who received at least one dose of CC-93538 and have any available concentration data. Only evaluable PK population was included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | CC-93538 360 mg QW | CC-93538 360 mg QW/Q2W
Number analyzed (Participants) | 110 | 97
ng/mL
  Pre-dose Week 24 | 148133.6 (69.9) | 151735.2 (55.8)
  Pre-dose Week 48: number analyzed (Participants) | 75 | 97
  Pre-dose Week 48 | 138545.4 (121.1) | 79884.3 (45.4)

ADVERSE EVENTS:
Time Frame: All Serious AEs, Non-Serious AEs and all cause mortality were collected from signing of informed consent form (Day -28) until 16 weeks after the last dose of CC-93538 or placebo was administered (Up to approximately 21 months).
Description: The Safety population consist of all randomized participants who received at least 1 dose of IP and analyzed based on the actual treatments they received.
Groups:
- CC-93538 360 mg Q2W: Participants with Eosinophilic Esophagitis received 360 mg CC-93538 SC once in a week (QW) in the 24-week induction phase and once every other week in 24-week maintenance phase.
Arm/Group | CC-93538 360 mg QW | CC-93538 360 mg Q2W | Placebo
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/117 | 0/143
Serious Adverse Events (participants affected / at risk) | 4/167 | 4/117 | 8/143
Other Adverse Events (participants affected / at risk) | 103/167 | 73/117 | 69/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CC-93538 360 mg QW (N=167) | CC-93538 360 mg Q2W (N=117) | Placebo (N=143)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Eosinophilic oesophagitis (Gastrointestinal disorders) | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Complication associated with device (General disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CC-93538 360 mg QW (N=167) | CC-93538 360 mg Q2W (N=117) | Placebo (N=143)
Abdominal pain (Gastrointestinal disorders) | 7 | 6 | 5
Diarrhoea (Gastrointestinal disorders) | 8 | 8 | 9
Nausea (Gastrointestinal disorders) | 11 | 6 | 6
Vomiting (Gastrointestinal disorders) | 6 | 10 | 4
Injection site reaction (General disorders) | 32 | 20 | 21
COVID-19 (Infections and infestations) | 29 | 28 | 21
Gastroenteritis (Infections and infestations) | 10 | 4 | 2
Influenza (Infections and infestations) | 3 | 6 | 4
Nasopharyngitis (Infections and infestations) | 16 | 14 | 13
Upper respiratory tract infection (Infections and infestations) | 17 | 11 | 12
Urinary tract infection (Infections and infestations) | 9 | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 9 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 6 | 4
Headache (Nervous system disorders) | 20 | 7 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT04753697/Prot_SAP_000.pdf